CLINICAL TRIAL: NCT00134849
Title: Hypertension in Management of Military Medicine
Status: Terminated | Type: Observational
Why Stopped: Inadequate number of records screened; primary investigator left institution.
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Other Study IDs: CIP #S-04-151
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a retrospective database review of primary care appointments of patients' charts with new diagnoses of hypertension.

DETAILED DESCRIPTION:
Compare the degree of blood pressure control of patients with stage 1 (BP < 130/80 mmHg) and stage 2 hypertension (BP > 20/10 mm Hg above goal BP) before and after the release of the Seventh report of Joint Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure (JNC 7) recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-09; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Maves, M.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States